CLINICAL TRIAL: NCT02427568
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Pilot Study of MDMA-Assisted Psychotherapy for Anxiety Associated With a Life-Threatening Illness
Brief Title: MDMA-Assisted Psychotherapy for Anxiety Associated With a Life-Threatening Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDA-1
Record Dates: First submitted 2015-04-13; First posted 2015-04-28 (Estimated); Results first posted 2021-08-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Anxiety
Keywords: Anxiety; MDMA; Life-threatening illness; Therapy; midomafetamine
MeSH Terms: conditions — Anxiety Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Placebo with therapy (Placebo Comparator): Inactive placebo administered on 2 blinded experimental sessions scheduled 2 to 4 weeks apart. Initial dose possibly followed 1.5 to 2.5 hours later by (optional) inactive placebo supplemental dose.
  Interventions: Drug: Placebo; Behavioral: Therapy
- MDMA-assisted therapy (125 mg) (Experimental): 125 mg midomafetamine HCl administered on 2 blinded experimental sessions scheduled 2 to 4 weeks apart. Initial dose possibly followed 1.5 to 2.5 hours later by a (optional) supplemental dose of 62.5 mg.
  Interventions: Drug: Midomafetamine HCl; Behavioral: Therapy

INTERVENTIONS:
Drug: Midomafetamine HCl — Two sessions of MDMA-assisted therapy lasting six to eight hours, scheduled two to four weeks apart.
  Other Names: 3,4-methylenedioxymethamphetamine; Midomafetamine; MDMA
  Arms: MDMA-assisted therapy (125 mg)
Drug: Placebo — Two sessions of placebo with therapy lasting six to eight hours, scheduled two to four weeks apart.
  Other Names: Inactive placebo
  Arms: Placebo with therapy
Behavioral: Therapy — Manualized therapy

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is safe and effective in people with anxiety associated with a life-threatening illness. The main question it aims to answer is: Does anxiety decrease in people receiving two sessions of MDMA-assisted therapy?

Researchers will compare people receiving placebo with therapy to people receiving MDMA-assisted therapy.

* Participants will undergo three non-drug preparatory therapy sessions before their first blinded session of MDMA or placebo with therapy.
* Each medication session will be followed by three non-drug integrative therapy sessions.
* After the second blinded medication session, participants receiving MDMA will complete a third open-label medication session.
* Participants who received placebo will be given the option to crossover and receive three sessions of assisted therapy.

DETAILED DESCRIPTION:
This Phase 2 pilot study is a randomized, double-blind, placebo-controlled study in 18 participants comparing the effects of MDMA-assisted therapy vs. placebo with therapy. Thirteen participants were randomized to the active dose condition of 125 mg of MDMA HCl (plus an optional supplemental dose of 62.5 mg MDMA HCl) with therapy and five participants were randomized to the placebo with therapy condition. The study consisted of two blinded experimental sessions of MDMA-assisted therapy or placebo with therapy, each session lasting six to eight hours and scheduled two to four weeks apart. Each participant was unblinded one month after their second experimental session in Stage 1. After unblinding, participants receiving MDMA were to complete a third open-label experimental session of MDMA-assisted therapy and participants who originally received placebo had the opportunity to cross over to open-label Stage 2 and receive active MDMA-assisted therapy in 3 sessions.

The primary objective of the study is to assess changes in trait anxiety in subjects receiving active dose MDMA compared to those receiving placebo as measured by State-Trait Anxiety Index (STAI) Trait scores from Baseline to the Primary Endpoint (one month after the second experimental session).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with life-threatening cancer or non-dementing neurological illness, which can be ongoing or in remission, but with a possibility of recurrence
* Prognosis of at least nine months life expectancy from the time of screening
* Have anxiety as a result of facing their illness
* Are at least 18 years old
* Are willing to refrain from taking any psychiatric medications during the study period;
* Are willing to commit to medication dosing, experimental sessions, follow-up sessions, and to complete evaluation instruments
* Are willing to remain overnight at the study site after each experimental session until after the integrative session occurring the next morning
* Must sign a medical release for the investigators to communicate directly with their therapist and doctors;
* Are willing to select up to three observers who will complete observer measures of subject attitudes and behavior
* Negative pregnancy test if able to bear children and agree to use effective birth control
* Are proficient in speaking and reading English
* Agree to have all psychotherapy sessions recorded to audio/video.

Exclusion Criteria:

* Are pregnant or nursing, or if a woman who can have children, those who are not practicing an effective means of birth control;
* Weigh less than 48 kg
* Are abusing illegal drugs
* Are unable to give adequate informed consent
* Upon review of past, current drugs/medication must not be on or have taken a medication that is exclusionary
* Upon review of medical or psychiatric history must not have any current or past diagnosis that would be considered a risk to participation in the study
* Have used "Ecstasy" (material represented as containing MDMA) at least once within twelve months of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wolfson, MD, Principal Investigator — Private Practice
Locations (1):
- Offices of Philip Wolfson MD, San Anselmo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share outcome data appearing in any published reports upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and study-related documents will be available when all participants have completed the study, and when data has been quality checked and locked.
Access Criteria: Interested persons should correspond with the central contact for the multisite study.

REFERENCES:
- [Result] Wolfson PE, Andries J, Feduccia AA, Jerome L, Wang JB, Williams E, Carlin SC, Sola E, Hamilton S, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. MDMA-assisted psychotherapy for treatment of anxiety and other psychological distress related to life-threatening illnesses: a randomized pilot study. Sci Rep. 2020 Nov 24;10(1):20442. doi: 10.1038/s41598-020-75706-1. PMID 33235285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through printed ads, internet ads, referrals from other psychiatrists, psychotherapists or physicians, and through word of mouth.
Groups:
- Placebo With Therapy: Inactive placebo administered on 2 blinded experimental sessions scheduled 2 to 4 weeks apart. Initial dose possibly followed 1.5 to 2.5 hours later by inactive placebo supplemental dose.
  Placebo with therapy: Two sessions of placebo with therapy lasting six to eight hours, scheduled two to four weeks apart.
- MDMA-assisted Therapy (125 mg): 125 mg midomafetamine HCl administered on 2 blinded experimental sessions scheduled 2 to 4 weeks apart. Initial dose possibly followed 1.5 to 2.5 hours later by a supplemental dose of 62.5 mg.
Period: Overall Study
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Started | 5 | 13
Completed | 5 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) set
Groups:
- MDMA-assisted Therapy (125 mg): 125 mg 3,4-methylenedioxymethamphetamine (MDMA) administered on 2 blinded experimental sessions scheduled 2 to 4 weeks apart. Initial dose possibly followed 1.5 to 2.5 hours later by a supplemental dose of 62.5 mg MDMA.
  MDMA-assisted therapy: Two sessions of MDMA-assisted therapy lasting six to eight hours, scheduled two to four weeks apart.
- Total: Total of all reporting groups
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg) | Total
Number analyzed (Participants) | 5 | 13 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (10.5) | 55.5 (7.0) | 54.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 3 | 12 | 15
  Race: Black/African American | 1 | 0 | 1
  Race: Other | 1 | 1 | 2
Baseline State-Trait Anxiety Inventory Trait (STAI-T) [Mean (Standard Deviation); unit: units on a scale] — The State-Trait Anxiety Inventory (STAI) Trait scale is a 20-item self-report measure of intensity of trait anxiety, defined as "long-standing nervous affect or anxiety disorder." Each item is rated on a 4-point scale ranging from 1 ('Not at all') to 4 ('Very Much So'). Items are summed for a total score ranging from 20 to 80, with higher scores indicating greater trait anxiety.
  units on a scale | 62.5 (7.31) | 57.4 (5.18) | 61.1 (7.03)

OUTCOME MEASURES:

1. Primary Outcome: Change in State Trait Anxiety Inventory (STAI) Trait Score From Baseline to Primary Endpoint
Description: The State-Trait Anxiety Inventory (STAI) is a 20-item self-report measure of intensity of anxiety. Each item consists of a 4-point Likert rating scale ranging from 1 ('Not at all') to 4 ('Very Much So'), with higher scores indicating greater anxiety. Items were summed for a total score that ranged from 20 to 80.
  The STAI differentiates between State Anxiety, defined as "anxiety experienced in reaction to a specific environmental circumstance," and Trait Anxiety, defined as "long-standing nervous affect or anxiety disorder." The use of the trait subscale as the primary outcome measure was intended to target those anxiety symptoms that are chronic and pervasive.
Time Frame: Baseline (3 months from enrollment) to Primary Endpoint (one month post-2nd experimental session)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale | -8.8 (14.7) | -23.5 (13.2)

2. Primary Outcome: Primary Endpoint STAI Trait Score
Description: The State-Trait Anxiety Inventory (STAI) is a 20-item self-report measure of intensity of anxiety. Each item consists of a 4-point Likert rating scale ranging from 1 ('Not at all') to 4 ('Very Much So'), with higher scores indicating greater anxiety. Items were summed for a total score that ranged from 20 to 80.
  The STAI differentiates between State Anxiety, defined as "anxiety experienced in reaction to a specific environmental circumstance," and Trait Anxiety, defined as "long-standing nervous affect or anxiety disorder." The use of the trait subscale as the primary outcome measure is intended to target those anxiety symptoms that are chronic and pervasive.
Time Frame: One month post-2nd experimental session
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale | 48.6 (12.6) | 38.9 (10.6)

3. Secondary Outcome: Change in STAI State Score From Baseline to Primary Endpoint
Description: The state subscale of the STAI (STAI-S) is a 20-item self-reported scale which assesses subjects' levels of transient, situationally oriented, anxiety. Like the trait subscale, participants respond to each item on the state subscale by selecting a response from a 4-point Likert scale ranging from 4 ("Not at all") to 1 ("Very much so"), with higher scores indicating greater anxiety. Items were summed for a total score that ranged from 20 to 80.
  The STAI differentiates between State Anxiety, defined as "anxiety experienced in reaction to a specific environmental circumstance," and Trait Anxiety, defined as "long-standing nervous affect or anxiety disorder." The use of the trait subscale as the primary outcome measure is intended to target those anxiety symptoms that are chronic and pervasive.
Time Frame: Baseline (3 months from enrollment) to Primary Endpoint (one month post-2nd experimental session)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale | -6.0 (15.8) | -22.1 (17.9)

4. Secondary Outcome: Change in Beck Depression Inventory-II (BDI-II) Score From Baseline to Primary Endpoint
Description: The Beck Depression Inventory-II (BDI-II) is a a 21-item self-reported measure of depression according to Diagnostic and Statistical Manual IV (DSM-IV) criteria. Each item is rated on a 4-point Likert scale ranging from 0 to 3. The total score is the sum of 21 items and range from 0 to 63. Score cutoffs indicate: 0-13 minimal depression, 14-19 mild depression, 20-28 moderate depression, and 29-63 severe depression. Higher scores indicate more severe depressive symptoms.
Time Frame: Baseline (3 months from enrollment) to Primary Endpoint (one month post-2nd experimental session)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale | -14.6 (8.6) | -20.9 (13.8)

5. Secondary Outcome: Change in Global Assessment of Functioning (GAF) Score From Baseline to Primary Endpoint
Description: The Global Assessment of Function (GAF) is a measure of a person's global social functioning made through clinical observation. The GAF consists of a single score, with scores ranging from 0 to 100, with 100 reflecting superior function and zero reflecting serious risk of causing harm to the self or others.
Time Frame: Baseline (3 months from enrollment) to Primary Endpoint (one month post 2nd experimental session)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale | 3.0 (12.5) | 6.6 (9.7)

6. Secondary Outcome: Change in MADRS Score From Baseline to Primary Endpoint
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item, clinician administered questionnaire used to diagnose the severity of depressive episodes. Each item has a score of 0 to 6. Overall scores are summed and range from 0 to 60. Score cutoffs indicate: 0-6 normal/symptom absent, 7-19 mild depression, 20-34 moderate depression, > 34 severe depression. Higher scores indicate greater severe depression.
Time Frame: Baseline (3 months from enrollment) to Primary Endpoint (one month post-2nd experimental session)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale | -7.0 (7.2) | -10.5 (8.2)

7. Secondary Outcome: Change in Pittsburgh Sleep Quality Inventory (PSQI) From Baseline to Primary Endpoint
Description: The Pittsburgh Sleep Quality Index (PSQI) is a measure of self-reported sleep quality over a one month period. It consists of 19 items with possible responses ranging from zero to four on a five-point scale. The PSQI consists of seven sub-scales: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medications, and daytime dysfunction. These are all summed to produce a single global scale. Global scores can range from 0 to 21, with higher scores reflecting poorer sleep quality, and a score below 5 indicating good sleep quality.
Time Frame: Baseline (3 months from enrollment) to Primary Endpoint (one month post-2nd experimental session)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale | -0.2 (1.3) | -3.6 (5.4)

8. Secondary Outcome: Change in Posttraumatic Growth Inventory (PTGI) From Baseline to Primary Endpoint
Description: The Posttraumatic Growth Inventory (PTGI) is a 21-item self-report measure of perceived growth or benefits occurring after a traumatic event. It contains five subscales; relationship to others, new possibilities, personal strength, spiritual change, and appreciation of life. Questions are answered on a scale from 0 (I did not experience this change) to 5 (I experienced this change to a great degree). Items are added to calculate the total PTGI score which ranges from 0 to 105, with higher scores indicative of greater growth.
Time Frame: Baseline (3 months from enrollment) to Primary Endpoint (one month post-2nd experimental session)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale | -2.6 (6.1) | 12.9 (23.2)

9. Secondary Outcome: Change in Functional Assessment of Chronic Illness Therapy Scale (FACIT) From Baseline to Primary Endpoint
Description: The Functional Assessment of Chronic Illness Therapy Scale (FACIT-Sp) is a 27-item self-report measure of quality of life issues specifically relevant to individuals with a chronic or life-threatening illness or condition. The core questionnaire consists of four subscales: Physical Well-being, Social/Family Well-being, Emotional Well-being, and Functional Well-being. Responses range from 0 (not at all) to 4 (very much), with higher scores indicating greater well-being. For each subscale, total scores were summed and range from 0 to 16.
Time Frame: Baseline (3 months from enrollment) to Primary Endpoint (one month post-2nd experimental session)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale
  Physical well-being | 2.8 (5.0) | 1.4 (4.4)
  Social/ family well-being | -2.0 (2.9) | 0.8 (3.4)
  Emotional well-being | 1.0 (2.2) | 1.6 (7.1)
  Functional well-being | 1.0 (1.6) | 4.8 (5.8)
  Additional concerns | -0.3 (5.0) | 4.5 (11.9)

10. Secondary Outcome: Change in Death Attitudes Profile (DAP) From Baseline to Primary Endpoint
Description: The Death Attitudes Profile (DAP) is a 32-item self-reported questionnaire that assesses individual attitudes and beliefs about death and dying. Each item on the scale is rated along a 7-point Likert scale ranging from "strongly disagree" (score of 1) to "strongly agree" (score of 7), with higher scores indicating more positive attitudes toward death.
  The DAP consists of 5 dimensions: fear of death (7 items summed with total scores ranging from 7 to 49), death avoidance (5 items summed with total scores ranging from 5 to 35), neutral acceptance (5 items summed with total scores ranging from 5 to 35), approach acceptance (10 items summed with total scores ranging from 10 to 70), and escape acceptance (5 items summed with total scores ranging from 5 to 35). For each dimension, a mean scale score can be computed by dividing the total scale score by the number of items forming each scale.
Time Frame: Baseline (3 months from enrollment) to Primary Endpoint (one month post-2nd experimental session)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale
  Fear of death | -0.6 (1.0) | -0.1 (0.6)
  Death avoidance | -1.1 (1.8) | 0 (0.8)
  Neutral acceptance | 0.2 (0.6) | 0.1 (0.6)
  Approach acceptance | -0.1 (1.1) | 0.3 (0.7)
  Escape acceptance | 0 (0.9) | 0.4 (1.0)

11. Secondary Outcome: Change in Self-Compassion Scale (SCS) From Baseline to Primary Endpoint
Description: The Self-Compassion Scale (SCS) is a 26-item self-reported questionnaire that assesses how respondents relate to themselves and treat themselves during difficult or painful experiences. Items are scored along a 5-point Likert-type scale ranging from 1 "almost never" to 5 "almost always." The SCS has six component (subscale) scores: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. Subscale scores are calculated by computing the mean of subscale item responses.
  A total self-compassion score is calculated by the sum of the subscale scores and range from 24 to 120 with higher scores indicating greater self compassion. Higher scores have been found to correlate with positive mental health outcomes, as well as decreased depression and anxiety.
Time Frame: Baseline (3 months from enrollment) to Primary Endpoint (one month post-2nd experimental session)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo With Therapy | MDMA-assisted Therapy (125 mg)
Number analyzed (Participants) | 5 | 13
score on a scale | -0.04 (0.5) | 0.4 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study: up to 2 months after the 2nd experimental session (for Stage 1 blinded for placebo group), at the end of Stage 1 (for MDMA group), up to 2 months after the 3rd experimental session (for Stage 2 crossover group), and at 12-month study follow-up (approximately 1 year following the 3rd MDMA session [following Stage 1 for participants in the MDMA arm and following crossover to Stage 2 for the Stage 1 placebo group] .
Groups:
- Placebo With Therapy (Blinded): Inactive placebo administered on 2 blinded experimental sessions scheduled 2 to 4 weeks apart. Initial dose possibly followed 1.5 to 2.5 hours later by (optional) inactive placebo supplemental dose.
  Placebo with therapy: Two sessions of placebo with therapy lasting six to eight hours, scheduled two to four weeks apart.
- MDMA-assisted Therapy (125 mg) (Blinded): 125 mg 3,4-methylenedioxymethamphetamine (MDMA) administered on 2 blinded experimental sessions scheduled 2 to 4 weeks apart. Initial dose possibly followed 1.5 to 2.5 hours later by a (optional) supplemental dose of 62.5 mg MDMA.
  MDMA-assisted therapy: Two sessions of MDMA-assisted therapy lasting six to eight hours, scheduled two to four weeks apart.
- Placebo Group Open-label Crossover to Unblinded MDMA-assisted Therapy (125 mg): Unblinded Crossover 125 mg 3,4-methylenedioxymethamphetamine (MDMA) administered on 3 open-label experimental sessions scheduled 2 to 4 weeks apart. Initial dose possibly followed 1.5 to 2.5 hours later by a (optional) supplemental dose of 62.5 mg MDMA.
- MDMA Group Open-label MDMA-assisted Therapy (125 mg): Open-Label 125 mg 3,4-methylenedioxymethamphetamine (MDMA) administered during open-label 1 experimental session. Initial dose possibly followed 1.5 to 2.5 hours later by a (optional) supplemental dose of 62.5 mg MDMA.
- Placebo With Therapy Group 12-month Follow-up: Follow-up with placebo with therapy group 12 months after end of Stage 2.
- MDMA-assisted Therapy Group 12-month Follow-up: Follow-up with MDMA-assisted therapy group 12 months after end of Stage 1.
Arm/Group | Placebo With Therapy (Blinded) | MDMA-assisted Therapy (125 mg) (Blinded) | Placebo Group Open-label Crossover to Unblinded MDMA-assisted Therapy (125 mg) | MDMA Group Open-label MDMA-assisted Therapy (125 mg) | Placebo With Therapy Group 12-month Follow-up | MDMA-assisted Therapy Group 12-month Follow-up
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/13 | 0/5 | 0/13 | 0/5 | 1/13
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/13 | 0/5 | 0/13 | 0/5 | 3/13
Other Adverse Events (participants affected / at risk) | 2/5 | 11/13 | 4/5 | 3/13 | 2/5 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo With Therapy (Blinded) (N=5) | MDMA-assisted Therapy (125 mg) (Blinded) (N=13) | Placebo Group Open-label Crossover to Unblinded MDMA-assisted Therapy (125 mg) (N=5) | MDMA Group Open-label MDMA-assisted Therapy (125 mg) (N=13) | Placebo With Therapy Group 12-month Follow-up (N=5) | MDMA-assisted Therapy Group 12-month Follow-up (N=13)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chordoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo With Therapy (Blinded) (N=5) | MDMA-assisted Therapy (125 mg) (Blinded) (N=13) | Placebo Group Open-label Crossover to Unblinded MDMA-assisted Therapy (125 mg) (N=5) | MDMA Group Open-label MDMA-assisted Therapy (125 mg) (N=13) | Placebo With Therapy Group 12-month Follow-up (N=5) | MDMA-assisted Therapy Group 12-month Follow-up (N=13)
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Balance Disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bruxism (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Clumsiness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dissociation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypomania (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 4 | 2 | 2 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Sinus Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tinea Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Muscle contractions (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-04-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT02427568/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT02427568/SAP_001.pdf
  • Informed Consent Form (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT02427568/ICF_002.pdf